CLINICAL TRIAL: NCT00718445
Title: Pennsylvania Consortium: Clinical Database
Status: Terminated | Type: Observational
Why Stopped: Terminated due to lack of funding and support staff
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-17445
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MND: * Patients seen in the MDA/ALS Center of Hope at Drexel University College of Medicine
  * Patients seen in the Department of Neurology at Drexel University College of Medicine

SUMMARY:
In order to streamline disease research in ALS and other motor neuron diseases, we have joined a consortium of clinical centers (Hershey and University of Pittsburgh) who will collaborate on clinical and basic research projects. As part of this collaboration, de-identified clinical data from subjects at each institution will be entered into a joint database kindly provided and maintained by the ALS Hope Foundation. This database is password protected and contains only de-identified information. In addition to clinical data, any research specimens that are available through IRB approved tissue collections will be linked to the subject so that the collaborating investigators can share samples and have the maximum information. This will enhance the usefulness of each specimen.

Once established, the database will provide a resource in which clinical data on a large number of patients along with tissue (blood, urine, muscle, csf, and autopsy) samples will be readily available. This will expedite research by circumventing the delays in collecting specimens prospectively and increase the number of specimens available by allowing the collaborating researchers access to each others specimens. In each case there will be a formal request placed to use specimens that are at the other institutions. These specimens will be used for research in the ALS Center of Hope at the Drexel University College of Medicine and shared with outside investigators with valid IRB approved protocols.

ELIGIBILITY:
Inclusion Criteria:

* Clinical data on patients with motor neuron diseases (ALS, PLS, Bulbar Palsy) and related disorders

Exclusion Criteria:

* Any patient without a motor neuron disease or related disorder

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the MDA/ALS Center of Hope at Drexel University College of Medicine Patients seen in the Department of Neurology at Drexel University College of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
None Specified | None Specified
  This database is intended to increase the efficiency of other IRB approved protocols by increasing accessibility of information and biological samples from the ALS cohort. No direct outcome measures have been specified for the creation of the database.

CONTACTS AND LOCATIONS:
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States